CLINICAL TRIAL: NCT04744519
Title: hCG Concentration in Peripheral Maternal Blood After Embryo Transfer, Ongoing Pregnancy
Brief Title: hCG Concentration in Peripheral Maternal Blood After Embryo Transfer, Ongoing Pregnancy Rates, and Morphokinetics
Status: Completed | Type: Observational
Sponsor: IVI Vigo (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 1712-VGO-122-EM
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: hCG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Collect data — - Controlled ovarian stimulation with GnRH antagonists effected to the patients in order to get their eggs through follicular puncture, which will be trigger by GnRH analogue. The eggs will be isolated and processed according to the standard protocol.
  Other Names: Collect retrospectively data on embryo implantation rate

SUMMARY:
hCG is a hormone produced very early by the embryo, but not by the oocyte. It has a pivotal role in the trophoblast differentiation, and embryo implantation as well as the corpus luteum support. In spite of its well-known role, the literature about it is scarce.

The aim of this retrospective study is to evaluate the relationship between the hCG concentration in peripheral maternal blood measured 11 days after embryo transfer, embryo morphokinetics pattern and the abortion and ongoing pregnancy rates.

We will study patients having transference of blastocyst cultured in time lapse monitored incubators and will check all the morphokinetics parameters with the IVI database.

DETAILED DESCRIPTION:
Human chorionic gonadotrophin is a two subunits (alpha and beta) glycoprotein hormone secreted by blastocyst trophoblastic cells.

It plays a role in progesterone secretion by corpus luteum, endometrium invasion and fusion by trophoectoderm, angiogenesis, and induction of trophoblast differentiation Shortly after embryo implantation, trophoblastic hCG is detectable in maternal blood, and its concetration depends on the number and functionality of trophoectoderm cells. Therefore, hCG concentration in maternal blood is measured as an early pregnancy marker.

However, hCG concentration in several women showed high variability, and embryo implantation also depends on endometrial receptivity, what means that in early stages, everything affecting endometrial receptivity, may affect hCG concentration.

Early high hCG concentration has been related with higher pregnancy rate and it has been proposed that hCG concentration may be related to the time of embryo implantation and the viable trophoectoderm cell number.

ELIGIBILITY:
Inclusion Criteria:

* Donors age < 32.
* IMC< 30kg/m2.
* Antral follicle count higher than 8.
* Single Blastocyst transference.
* 5% oxygen embryo culture,
* time-lapse monitoring incubation KID embryos.

Exclusion Criteria:

* Müllerian anomalies,
* Hydrosalpinx.
* Any indication of oocyte vitrification.
* Severe male factor.
* Embryos transferences where a tenaculum was required, or more than one attempt was needed.

Ages: 18 Years to 32 Years | Sex: Female
Age Groups: Adult
Study Population: Patients who underwent ICSI with oocyte donation in IVI Vigo under time-lapse monitoring between 2013 and up to June 2019.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Researchers pretend to correlate the quality of the trophoectoderm and the embryo morphokinetics time with the hCG concentration after 13 days of embryo transfer, and also the implantation and the ongoing pregnancy rate. | Since 2013 to april 2019
  • Clinical pregnancy: when the maternal serum levels of β-hCG are higher than 10 UI/L, between 14 and 16 days after the fertilization and the presence of a gestational sac can be appreciated by ultrasound scan a week later (21-23 days after fertilization)

CONTACTS AND LOCATIONS:
Overall Officials: Elkin Muñoz, Study Director — IVI Vigo
Locations (1):
- IVI Vigo, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basile N, Nogales Mdel C, Bronet F, Florensa M, Riqueiros M, Rodrigo L, Garcia-Velasco J, Meseguer M. Increasing the probability of selecting chromosomally normal embryos by time-lapse morphokinetics analysis. Fertil Steril. 2014 Mar;101(3):699-704. doi: 10.1016/j.fertnstert.2013.12.005. Epub 2014 Jan 11. PMID 24424365
- [Background] Dominguez F, Gadea B, Esteban FJ, Horcajadas JA, Pellicer A, Simon C. Comparative protein-profile analysis of implanted versus non-implanted human blastocysts. Hum Reprod. 2008 Sep;23(9):1993-2000. doi: 10.1093/humrep/den205. Epub 2008 Jun 12. PMID 18556682